CLINICAL TRIAL: NCT05792319
Title: Clinical Profile and Out Come of Children With Wilson's Disease :A Single Tertiary Center Study .
Brief Title: Clinical Profile and Out Come of Children With Wilson's Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rehab Ahmed Ali, Clinical profile and out come of Children with Wilson's disease, Assiut University
Other Study IDs: COC of WILSON disease
Record Dates: First submitted 2023-02-09; First posted 2023-03-31 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-11

CONDITIONS: Clinical Outcome in WILSON Disease
MeSH Terms: interventions — Urination; Liver Function Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 24 hour copper in urine and liver function test — sampling 24 hour copper in urine and liver function test

SUMMARY:
Clinical profile and out come of Children with Wilson's disease :A single tertiary center study

DETAILED DESCRIPTION:
Wilson disease (WD) is an autosomal-recessive disorder of copper metabolism caused by mutations in the ATP7B gene . It presents in childhood, adolescence or adulthood with a wide range of clinical manifestations. The disease prevalence has previously been estimated as 1 in 30,000 , but some recent analyses have suggested a genetic prevalence of 1 in 7,000 . Copper is absorbed from the stomach and duodenum, taken up by the liver, and secreted by the liver into the systemic circulation bound to ceruloplasmin ATP7B transports copper through the trans-Golgi network in hepatocytes before it is incorporated into apoceruloplasmin which is secreted as holoceruloplasmin.

ATP7B is also essential for biliary excretion of copper when cytoplasmic levels are high. Dysfunction of ATP7B therefore leads to accumulation of copper in the liver giving rise to cellular damage and disease, and the release of nonceruloplasmin bound copper into the systemic circulation. Copper also accumulates and is associated with cellular damage and disease in other organs mostly in the brain Typical presentation of WD is in adolescence to early adulthood, but it may occur at any age . Clinical presentation can vary widely in terms of type and severity, but the key features are various degrees of liver disease,

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 1-18 years
* fulfill the criteria for diagnosis of Wilson's disease according to Wilson's score

Exclusion Criteria:

1. persistent neonatal jaundice.
2. Patients presented with Acute and chronic liver disease rather than Wilson's e.g

   1. Autoimmune hepatitis
   2. Hepatitis C virus ,
   3. Hepatitis B virus infection ,(d)Hepatic focal lesions and(e) Metabolic liver disease e.g Gauchier ,glycogen storage disease and Niemman pick .

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The aim of this study to describe the clinical profile of children diagnosed as Wilson's disease who were admitted to A.U.C.H and explore the out come of these patients either they receive the chelation therapy or not along a period of one year
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
COC in WILSON disease | Baseline
  Clinical profile and out come of Children with Wilson's disease :A single tertiary center study

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tryambak S, Sumanta L, Radheshyam P, Sutapa G. Clinical profile, prognostic indicators and outcome of Wilson's disease in children: a hospital based study. Trop Gastroenterol. 2009 Jul-Sep;30(3):163-6. PMID 20306753